CLINICAL TRIAL: NCT05880316
Title: Prevalence of Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD) Among Nurses in a Single Tertiary Care Centre and the Role of Intermittent Fasting in Improving Hepatic Steatosis
Brief Title: Prevalence of MAFLD Among Nurses and the Role of Intermittent Fasting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Khairul Najmi, Dr, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKM/PPI/111/8/JEP-2023-276
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Fatty Liver Disease
Keywords: fatty liver; MAFLD; intermittent fasting; transient elastography; fibroscan
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting Group (Experimental): IF regime: 3 fasting day: 4 non-fasting day. On fasting day - allows to eat restricted calorie diet (up to 70% total daily calorie intake) for 8 hours.
  Interventions: Behavioral: Intermittent Fasting
- Non-Fasting Group (No Intervention): Usual care. Not allowed to fast

INTERVENTIONS:
Behavioral: Intermittent Fasting — 3:4 regime
  Arms: Intermittent Fasting Group

SUMMARY:
This study consists of 2 parts:

Part 1: a cross-sectional study, looking at the prevalence of metabolic dysfunction-associated fatty liver disease (MAFLD) among nurses in Hospital Canselor Tuanku Muhriz (HCTM).

Part 2: a randomized controlled trial of intermittent fasting with MAFLD subjects.

DETAILED DESCRIPTION:
The investigators aim to screen at least 350 participants for fibroscan-detected fatty liver. Baseline anthropometric data will be taken. Questionnaires on dietary habits - Foof Frequency Questionnaire (FFQ) and exercise habits - International Physical Activity Questionnaire (IPAQ) will be done.

Approximately 100 participants who have fatty liver from Part 1 study, will be enrolled and randomized into Part 2. The intervention group will undergo intermittent fasting (3 fasting day:4 non-fasting days) while the control group will continue the usual standard care, for 8 weeks.

Measurements pre- and post-intervention include Fibroscan measurement, blood LiverFASt, anthropometric data, and exercise habit (IPAQ).

ELIGIBILITY:
Inclusion Criteria:

* nurses at HCTM, 18 years and above

Exclusion Criteria:

* pregnancy
* previous bariatric surgery
* liver cirrhosis
* liver cancer
* steatogenic drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-28 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean change of controlled attenuated parameter (CAP) (dB/m) | 8 weeks
  hepatic steatosis score - measured by transient elastography (Fibroscan). The higher the value, the more severe the degree of steatosis. Range of score: 100-500dB/m

SECONDARY OUTCOMES:
Mean change of hepatic fibrosis score (kPa) | 8 weeks
  measured by transient elastography (Fibroscan). The higher the value, the more severe the degree of fibrosis. Range of score: 1-25 kPa
Mean change of steatotest, actitest, and fibrotest scores | 8 weeks
  measured by blood test LiverFASt. The higher the value, more severe the degree of steatosis, inflammation, and fibrosis. Range of score: 0 - 1
mean change of Body Mass Index | 8 weeks
  The higher the value, the more overweight/obese patient is. BMI is measured by (weight in kg/height x height in meter). BMI category is based on Asian classification: <18.5: underweight, 18.5 - 22.9: normal, 23 - 27.5: overweight, >27.5 obese

CONTACTS AND LOCATIONS:
Overall Officials: Khairul Najmi M Nawawi, Principal Investigator — Gastroenterology Unit, Department of Medicine, Faculty of Medicine, UKM
Locations (1):
- Hospital Canselor Tuanku Muhriz, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
undecided